CLINICAL TRIAL: NCT03385746
Title: Evaluation of Retention of Metal Reinforced Polyamide Denture Base Compared to Conventional Heat Cured Acrylic Resin Denture Base in Complete Mandibular Denture
Brief Title: Retention of Metal Reinforced Polyamide Denture Base and Heat Cured Acrylic Resin Denture Base in Complete Mandibular Denture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Hassan, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: re inforced complete denture
Record Dates: First submitted 2017-12-21; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Anodontia of Permanent Dentition
MeSH Terms: conditions — Anodontia of Permanent Dentition | interventions — Nylons

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polyamide (Experimental): metal reinforced polyamide denture base material
  Interventions: Other: polyamide
- heat cured acrylic resin (Active Comparator): conventional heat cured acrylic resin denture base
  Interventions: Other: heat cured acrylic resin

INTERVENTIONS:
Other: polyamide — metal reinforced polyamide denture base material
  Other Names: Nylon
  Arms: polyamide
Other: heat cured acrylic resin — conventional heat cured acrylic resin denture base material
  Arms: heat cured acrylic resin

SUMMARY:
The trial is done in order to reinforce polyamide to improve its modulus of elasticity to be able to use it as a denture base material in all clinical cases

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with age range from fifty five to sixty five completely edentulous and in good medical condition
2. Patients have skeletal Angle's class I maxillo-mandibular relationship and sufficient inter arch distance.
3. Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
4. Free from any tempro-mandibular disease.
5. Good oral hygiene.

Exclusion Criteria:

1. Neuromuscular disorder and orofacial disease.
2. Tempromandibular joint and muscle pain
3. xerostomia or excessive salivation.
4. Limited mouth opening

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Retention assessed by digital forcemeter | 6 weeks
  Retention of mandibular denture

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vojdani M, Giti R. Polyamide as a Denture Base Material: A Literature Review. J Dent (Shiraz). 2015 Mar;16(1 Suppl):1-9. PMID 26106628
- [Background] Soygun K, Bolayir G, Boztug A. Mechanical and thermal properties of polyamide versus reinforced PMMA denture base materials. J Adv Prosthodont. 2013 May;5(2):153-60. doi: 10.4047/jap.2013.5.2.153. Epub 2013 May 30. PMID 23755341